CLINICAL TRIAL: NCT00086073
Title: Parkinson's Disease Collaborative Study of Genetic Linkage
Brief Title: Parkinson's Research: The Organized Genetics Initiative
Acronym: PROGENI
Status: Completed | Type: Observational
Sponsor: Indiana University School of Medicine (Other)
Collaborators: The Parkinson Study Group (Network); Children's Hospital Medical Center, Cincinnati (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Tatiana Foroud, Ph.D, Principal Investigator, Indiana University
Organization: Indiana University (Other)
Other Study IDs: 9703-09; R01NS037167 (NIH)
Record Dates: First submitted 2004-06-22; First posted 2004-06-24 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2010-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Parkinson's disease; PD; genetics; genes; siblings; family
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this trial is to study genetic and other risk factors that may be important in the development of Parkinson's disease.

DETAILED DESCRIPTION:
The The Parkinson's Research: The Organized Genetics Initiative, also known as PROGENI, is a multi-center study involving 2000 people throughout North America who are affected, or possibly affected, with Parkinson's disease (PD). The goal of the initiative is to study the genetic and other risk factors which may be important in the development of PD.

In order to better understand the genetic factors leading to PD, researchers will study families having 2 or more members diagnosed with PD. Using DNA samples from each participant, researchers hope to identify genes that may cause a person to be at higher risk for developing PD.

Each participant in the study will be asked to complete a family history questionnaire, providing information about the history of PD in the family. Participants also will be asked to discuss the symptoms they have experienced and their responses to PD medications. This information will be used by study personnel to determine further eligibility for the study. Those eligible for further participation will be asked to undergo a study visit at the site closest to their residence, during which they will be asked to complete questionnaires regarding PD symptoms, medical history, places of residence, occupations, mood, mental status, and activity level. A blood sample will be drawn for DNA extraction. The study visit will take about 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study participants must be diagnosed with or have symptoms of PD. In addition, they must also have a family history of PD in other relatives.

Exclusion Criteria:

* Subjects cannot have participated in any other genetic research project for Parkinson's disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: families having 2 or more members diagnosed with PD
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 1998-08; Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Foroud, Ph.D., Principal Investigator — Indiana University
Locations (57):
- United States (51):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Parkinson's & Movement Disorder Institute, Fountain Valley, California
  - University of California Irvine, Irvine, California
  - Pacific Neuroscience Medical Group, Inc, Oxnard, California
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Colorado Neurological Institute, Englewood, Colorado
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Parkinson's Disease & Mmvt Disorders Ctr of Boca Raton, Boca Raton, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Pacific Health Research Institute, Honolulu, Hawaii
  - Northwestern University Medical School, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Southern Illinois Univ School of Medicine, Springfield, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Oschsner Clinic Foundation, New Orleans, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Port City Neurology, Inc, Scarborough, Maine
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Henry Ford Health System, Southfield, Michigan
  - University of Minnesota Fairview Univ Med Ctr, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - University of Buffalo, Buffalo, New York
  - Beth Israel Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia-Presbyterian Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Medical College of Ohio, ,, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburg, Pittsburgh, Pennsylvania
  - Neurohealth, Warwick, Rhode Island
  - University of Tennessee-Health Sciences Center, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - London Health Sciences Center, London, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Hotel-Dieu Hospital-CHUM, Montreal, Quebec
- University of Puerto Rico School of Medicine, San Juan, Puerto Rico